CLINICAL TRIAL: NCT02387645
Title: LUDEC Study - Pilot Study of the Lavage of the Uterine Cavity for the Diagnosis of Endometrial Carcinoma
Acronym: LUDEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Paul Speiser, Prof.MD,, Professor Dr. (M.D.), Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EK1237/2014
Record Dates: First submitted 2015-03-08; First posted 2015-03-13 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Cancer of Endometrium; Carcinoma of Endometrium; Endometrial Neoplasms
Keywords: Endometrium; Endometrial Neoplasms; Early detection; Carcinoma of Endometrium; Gynaecological Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients prior to surgery for EC/suspicion (Experimental): Patient undergoing surgery for strong suspicion of EC
  Interventions: Procedure: Lavage of the Uterus

INTERVENTIONS:
Procedure: Lavage of the Uterus — The lavage will be performed in the operating theatre under general anesthesia. The ALPINE technique includes the following steps. A three way catheter (catheter for uterine and tubal lavage) is inserted into the cervical canal and a balloon is inflated to seal the cervical canal. The patient is put into anti-Trendellenburg positioning. Normal saline is slowly flushed into the uterine cavity and proximal tubes. After the lavage is finished, the balloon is deflated and the catheter is removed. A cap is put on the collection syringe and the syringe is sent to the laboratory.

SUMMARY:
The current pilot study aims at answering the scientific question, whether exfoliated cells from Endometrium Carcinoma (EC) can be detected in the lavage fluid from the uterine cavity and proximal fallopian tubes with the same sensitivity as in specimen from liquid-based cervical cytology. If this turns out to be the case, earlier detection, particularly of type II EC should be possible.

DETAILED DESCRIPTION:
Endometrial Carcinoma (EC) - carcinoma of the lining of the uterus - is the most common gynecologic malignancy in western civilized countries. Just in the US, approximately 42,160 cases are diagnosed and 7,780 deaths occur annually.

Type I EC is estrogen-dependent and associated with conditions that elevate estrogen levels. The precursor lesion, atypical endometrial hyperplasia, is well described. Type I EC, often of endometroid histology, well differentiated in most cases, is usually diagnosed at an early stage due to irregular bleeding and therefore has a good prognosis.

Type II EC is not estrogen-dependent and of serous or clear cell histology. In contrast to type I cancers, the vast majority, especially of serous cancers, are high grade, affect postmenopausal women, do not cause early symptoms, are diagnosed at an advanced stage, behave more like epithelial ovarian cancer (EOC) and have a very poor prognosis. Precursor lesions in the endometrium are referred to as "serous endometrial intraepithelial carcinoma" (SEIC), lesions quite similar to the precursor lesion of EOC in the fallopian tube, called "serous tubal intraepithelial carcinoma" (STIC).

Unfortunately, most patients with type II epithelial EC, in particular the serous and clear cell carcinomas, experience few or no symptoms until the disease has metastasized. The lack of early symptoms and the absence of a reliable screening test to detect the disease early, result in women being diagnosed after the disease has spread beyond the uterus and therefore has a poor prognosis. For these reasons, there is a clear medical need for earlier diagnosis of type II EC.

Type I and type II uterine tumors also appear to have a different pattern of molecular alterations that underlie pathogenesis and/or progression (1). Alterations in the tumor suppressor gene PTEN, microsatellite instability, and K-ras alterations have been associated with the early development of type I tumors, while these alterations are uncommon in type II cancers. On the other hand, mutations in the TP53 gene appear to be important in the early pathogenesis of uterine serous carcinomas. Moreover, HER2 overexpression/amplification has been associated with type II tumors.

Irregular bleeding as the main symptom of EC is conventionally investigated by "dilation and curettage" and hysteroscopy, a rather invasive procedure requiring general anesthesia and hospital admission. This allows for diagnosis of early stage type I and usually endometroid carcinoma. Bleeding from serous type II EC is examined the same way, but usually, the disease has already progressed into an advanced stage at the time of diagnosis.

The proof of concept that malignant cells from the upper genital tract get transported even into the lower genital tract was recently published by Kinde I. et al. (2). Liquid-based cervical cytology allows not only cytological evaluation but also collection of DNA. A panel of genes that are commonly mutated in endometrial and ovarian cancers was assembled with new whole-exome sequencing data from 22 endometrial cancers and previously published data on other tumor types, including mutations in the TP53 gene. This panel was used to search for mutations in 24 endometrial and 22 ovarian cancers and identified mutations in all 46 samples. Aiming at establishing a possible screening test for EOC and EC, tumor cells were searched for in the DNA obtained through liquid Pap smear. With a sensitive massively parallel sequencing method, it was possible to identify the same mutations in the DNA from liquid Pap smear specimens in 100% of endometrial cancers (24 of 24) and in 41% of ovarian cancers (9 of 22).

A promising approach for the detection of EOC has been established by Paul Speiser and Robert Zeillinger (Molecular Oncology Group, Department of General Gynaecology and Gynaecologic Oncology, Medical University of Vienna, Austria). This approach is called the ALPINE technique (Austrian Lavage Procedure for the Detection of tubal Intraepithelial Neoplasms) (manuscript under preparation). It includes a lavage of the uterine cavity and proximal fallopian tubes and subsequent analysis of this lavage fluid for the presence of pre-malignant and malignant cells.

Uterine lavages were collected before a surgical intervention for suspected ovarian malignancy at the investigators' institution. After malignancy was confirmed, a panel of genetic changes frequently found in endometrial and ovarian cancers (see below) were studied in the lavage samples of 22 ovarian carcinoma patients through deep sequencing by the group of Bert Vogelstein (Johns Hopkins University, Baltimore, USA). The presence of genetic changes, indicative for ovarian cancer, could be confirmed in 16/22 (~73%) lavage specimen.

The sensitivity in detecting EOC in this pilot study is unprecedented and has sparked further studies, examining the potential of the ALPINE technique in detecting EOC and the precursor lesion of EOC, called STIC. The fact that ovarian cancer cells - collected through the ALPINE technique - were detected with a much higher sensitivity in the lavage, compared to liquid-based cervical cytology, makes the investigators confident that EC detection in lavage specimen should also be possible. If it turns out that already SEICs can be detected in the lavage specimen, this could even result in prevention of type II EC.

The investigators will study about 80 lavage samples and the corresponding EC tissue samples in women who undergo "dilation and curettage" and hysteroscopy for abnormal uterine bleeding and suspected EC. Women who were diagnosed with EC and are scheduled for hysterectomy can also be included in the study. Patients will be recruited into the study until 40 cases of verified ECs and corresponding lavages are collected.

Before "dilation and curettage" and hysteroscopy for abnormal uterine bleeding or before hysterectomy for EC, a lavage of the uterine cavity and proximal fallopian tubes will be obtained. The lavage will be performed in the operating theatre under general anesthesia.

After the lavage is finished, a cap is put on the collection syringe and the syringe is sent to the laboratory. The 10ml uterine aspirate will be centrifuged for 10 minutes at 300 x g. The supernatant and the remaining cell pellet will be frozen at -80°C.

Analysis of the cell pellet will be carried out applying the sensitive massively parallel sequencing method published by Kinde et al. (2). Mutations in the following genes will be analysed: AKT1, APC, BRAF, CTNNB1, EGFR, FBXW7, KRAS, NRAS, PTEN, PIK3CA, PPP2R1A, and TP53.

Considerations on safety and ethical issues:

One concern with the lavage procedure might be that tumor cells from EC might get washed into the peritoneal cavity during the procedure.

During hysteroscopy, the distention media drains through the tubes into the peritoneal cavity in large quantities. A meta-analysis of observational studies reported no significant difference in the frequency of positive peritoneal cytology in women with EC who had or had not undergone diagnostic hysteroscopy (3).

This indicates that transport of EC cells from the uterine cavity into the peritoneal cavity during diagnostic hysteroscopy does not necessarily result in implantation and persistence. In the few studies that have reported long-term follow-up, there was no detriment to survival associated with pre-staging hysterosalpingography (with confirmed intraperitoneal spill) (4) or hysteroscopy (5).

These findings are very reassuring that the lavage of the uterine cavity and proximal tubes by the ALPINE technique is safe.

Conclusion:

If it is possible to detect EC with a very high sensitivity and specifisity by mutation analysis in the lavage of the uterine cavity and fallopian tubes, this result will represent an important finding and might open the opportunity for earlier detection of EC, possibly resulting into a stage shift to earlier stages. That would lead to an improvement of the prognosis, even in type II EC.

Literature:

1. Lax SF Molecular genetic pathways in various types of endometrial carcinoma: from a phenotypical to a molecular-based classification. Virchows Arch. 2004;444(3):213.
2. Kinde I et al. Evaluation of DNA from the Papanicolaou Test to Detect Ovarian and Endometrial Cancers. Sci Transl Med. 2013 Jan 9;5(167):167ra4
3. Yazbeck C, Dhainaut C, Batallan A, et al. [Diagnostic hysteroscopy and risk of peritoneal dissemination of tumor cells]. Gynecol Obstet Fertil 2005; 33:247.
4. Devore GR, Schwartz PE, Morris JM. Hysterography: a 5-year follow-up in patients with endometrial carcinoma. Obstet Gynecol 1982; 60:369.
5. Ben-Arie A, Tamir S, Dubnik S, et al. Does hysteroscopy affect prognosis in apparent early-stage endometrial cancer? Int J Gynecol Cancer 2008; 18:813.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing "dilation and curettage" and hysteroscopy for abnormal uterine bleeding
* Patients undergoing hysterectomy for EC

Exclusion Criteria:

* pregnant
* incapacitated persons

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Detection of EC with a very high sensitivity and specifisity - by mutation analysis of cell material gained through the lavage of the uterine cavity and fallopian tubes. | 10 minutes
  preoperative

CONTACTS AND LOCATIONS:
Overall Officials: Paul Speiser, Prof. Dr. med., Study Chair — Medical University Vienna, Dptm. of Obstetrics & Gynaecology; Elisabeth Maritschnegg, MSc., Study Chair — Medical University Vienna, Dptm. of Obstetrics & Gynaecology
Locations (1):
- Medical University Vienna, Dptm. of Obstetrics & Gynaecology, Vienna, Austria